CLINICAL TRIAL: NCT07019779
Title: A Multicenter, Open-Label, Phase I/II Clinical Study to Evaluate CM518D1 in the Treatment of Patients With Advanced Solid Tumors
Brief Title: Study of CM518D1 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM518D1-030101
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase I dose escalation (Experimental)
  Interventions: Biological: CM518D1
- Phase I dose expansion (Experimental)
  Interventions: Biological: CM518D1
- Phase II (Experimental)
  Interventions: Biological: CM518D1

INTERVENTIONS:
Biological: CM518D1 — CM518D1 will be administered intravenously once every 3 weeks (Q3W) in 6 predetermined dose levels.
  Arms: Phase I dose escalation
Biological: CM518D1 — CM518D1 will be administered intravenously once every 3 weeks (Q3W) in one or more potential recommended phase 2 dose(RP2D).
  Arms: Phase I dose expansion
Biological: CM518D1 — CM518D1 will be administered intravenously once every 3 weeks (Q3W) in different types of solid tumor cohorts.
  Arms: Phase II

SUMMARY:
This is an interventional study to assess the safety, tolerability, efficacy, pharmacokinetics, and immunogenicity of CM518D1 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female ≥ 18 and ≤75 years of age.
* 2. Subjects with histologically or cytologically confirmed advanced solid tumors.
* 3. At least one measurable lesion according to RECIST v1.1.
* 4. Expected survival time ≥ 3 months as judged by the Investigator.

Exclusion Criteria:

* 1. Subjects who have received any chemotherapy or any drug therapy for antitumor treatment including monoclonal antibodies, targeted therapy, radioimmunoconjugates, or Antibody-Drug Conjugates(ADCs), or any investigational product therapy for anti-tumor therapy within 28 days prior to the first dose or within 5 half-lives (whichever is shorter).
* 2. Subjects who have received major surgery within 28 days prior to the first dose.
* 3. Subjects who have received radiotherapy within 21 days prior to the first dose.
* 4. Subjects who have received systemic glucocorticoid therapy (more than 10 mg of prednisone or equivalent daily) or other forms of immunosuppressive therapy within 7 days prior to the first dose.
* 5. Subjects who have received any CDH17-targeted therapy.
* 6. History of other malignancies within 5 years prior to the first dose, excluding cured basal or squamous cell carcinoma of skin, carcinoma cervix in situ, or breast ductal carcinoma in situ.
* 7. Hypersensitivity to the investigational drug or its excipients.
* 8. Pregnant or lactating female patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT)-Phase I dose escalation | First cycle (21 days)
  DLT is defined as a toxicity occurring during the DLT observation period.
Incidence of adverse events (AEs), serious adverse events (SAEs), and specific laboratory abnormalities-Phase I dose escalation | Through study completion, an average of 2 years.
  An adverse event is defined as any unfavorable medical event that occurs in a subject after receiving the investigational drug, which will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria.
Incidence of adverse events (AEs), serious adverse events (SAEs), and specific laboratory abnormalities-Phase I dose expansion | Through study completion, an average of 2 years.]
  An adverse event is defined as any unfavorable medical event that occurs in a subject after receiving the investigational drug, which will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria.
Preliminary efficacy-Phase I dose expansion | Through study completion, an average of 2 years.]
  Preliminary efficacy includes objective response rate (ORR), duration of response (DOR), disease control rate (DCR), time to response (TTR), and progression-free survival (PFS).
Objective response rate (ORR)-Phase II | Through study completion, an average of 2 years.]
  ORR is defined as the proportions of subjects with a complete response (CR) and partial response (PR). ORR will be assessed by investigator according to Response Evaluation Criteria in Solid Tumors( RECIST) v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center (SYSUCC), Guangzhou, Guangdong, China